CLINICAL TRIAL: NCT04550325
Title: A Phase 1/2 Open Label, Multicenter, Single Arm Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Single Dose Kamada Anti-SARS-CoV-2 in COVID-19 Hospitalized Patients With Pneumonia
Brief Title: Safety, PK and PD of Kamada Anti-SARS-CoV-2 in COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kamada Anti-SARS-CoV-2-001
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Pneumonia, Viral
MeSH Terms: conditions — COVID-19; Pneumonia, Viral

STUDY DESIGN:
Intervention Model Description: A Phase 1/2 Open Label, Single Arm Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Single Dose Kamada Anti-SARS-CoV-2 in COVID-19 Hospitalized Patients with Pneumonia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immune gamma globulin (IgG) (Experimental): Single dose of 4g Immune gamma globulin (IgG) preparation Kamada Anti-SARS-CoV-2 given as an intravenous infusion
  Interventions: Biological: Kamada Anti-SARS-CoV-2

INTERVENTIONS:
Biological: Kamada Anti-SARS-CoV-2 — Anti-SARS-CoV-2 is a preparation of immune gamma globulin manufactured from convalescent plasma of COVID-19 recovered patients, using Kamada's proprietary purification methods

SUMMARY:
Evaluate the safety pharmacokinetics and pharmacodynamics (PK/PD)of a single dose of Kamada anti-severe acute respiratory syndrome (SARS)- CoV-2 in patients hospitalized with COVID-19 caused pneumonia

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Laboratory confirmed SARS-CoV-2 infection by nasopharyngeal swab Real time polymerase chain reaction (RT-PCR)
3. Hospitalized for COVID-19 pneumonia
4. Dosing should be within 10 days of symptom start
5. Able and willing to sign informed consent form

Exclusion Criteria:

1. History of hypersensitivity to plasma products and/or severe Immunoglobulin A deficiency (< 7 mg/dL)
2. Requirement of high flow oxygen devices, or non-invasive ventilation or mechanical ventilation, or extracorporeal membrane oxygenation (ECMO) at screening
3. Cardiovascular instability
4. History of thrombo-embolic events
5. Acute renal failure or creatinine >2 mg/dL or estimated estimated glomerular filtration rate (eGFR) <30 mL/min
6. History of lung transplantation
7. Major surgery (abdominal and chest) within the last 4 weeks
8. Severe chronic background disease, per investigator's judgement for example, Cirrhosis grade C, Dialysis, cardiac insufficiency (NYHA III), pulmonary disease (FEV1<50 percent of predicted) etc.
9. Pregnancy or lactation
10. Treatment with plasma units or immunoglobulin preparations within the last 4 weeks
11. Participation in another pharmaceutical interventional clinical study within 4 weeks from screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Adverse events, serious adverse events, and deaths | 14 days
  Record adverse events, serious adverse events, and deaths
Adverse events, serious adverse events, and deaths | 28 days
  Record adverse events, serious adverse events, and deaths

SECONDARY OUTCOMES:
AUC0-7 of Anti SARS CoV-2 antibodies | 7 days
  Measurement of the area under the curve of anti SARS CoV-2 immunoglobulin
Neutralization activity | 7 days
  Evaluate virus neutralization activity of patient's plasma

OTHER OUTCOMES:
Duration of Hospitalization | 84 days
  Time patient spent in hospital
Clinical status on the 6 point ordinate scale | 84 days
  Score on the 6 point ordinate scale

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center Hospital- Tel Hashomer, Ramat Gan
  - Kaplan Medical Center, Rehovot